CLINICAL TRIAL: NCT04460066
Title: A Randomized, Double-blind, Placebo-controlled Phase Ib/II Clinical Study of Anti-pd-l1 Monoclonal Antibody Injection (ZKAB001) Combined Albumin Binding Paclitaxel, Cisplatin in Neoadjuvant Treatment of Esophageal Squamous Cell Carcinoma.
Brief Title: A Study of Anti-PD-L1 Antibody in Neoadjuvant Chemotherapy of Esophageal Squamous Cell Carcinoma.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKAB001-LEES-2020-02
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Albumin-Bound Paclitaxel; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-L1 group (Experimental): All patients will receive 16 cycles of anti-PD-L1 antibody (5mg/kg, IV, every 3 weeks) , concurrently with 4 cycles of albumin-bound paclitaxel and cisplatin (albumin-bound paclitaxel 125mg/m2 on days 1, 8 and cisplatin 75 mg/m2 on day 1 every 3 weeks).
  Interventions: Drug: anti-PD-L1 antibody; Drug: albumin bound paclitaxel; Drug: cisplatin; Procedure: radical resection of esophageal carcinoma
- placebo group (Placebo Comparator): All patients will receive 4 cycles of placebo ( IV, every 3 weeks) , concurrently with 4 cycles of albumin-bound paclitaxel and cisplatin (albumin-bound paclitaxel 125mg/m2 on days 1, 8 and cisplatin 75 mg/m2 on day 1 every 3 weeks).
  Interventions: Drug: albumin bound paclitaxel; Drug: cisplatin; Drug: placebo; Procedure: radical resection of esophageal carcinoma

INTERVENTIONS:
Drug: anti-PD-L1 antibody — Patients will receive 16 cycles of anti-PD-L1 antibody 5mg/kg IV on day 1 every 3 weeks.
  Other Names: ZKAB001; Socazolimab Injection
  Arms: PD-L1 group
Drug: albumin bound paclitaxel — Patients will receive 4 cycles of albumin bound paclitaxel 125mg/m2 on days 1, 8 every 3 weeks .
  Other Names: ABRAXANE
Drug: cisplatin — Patients will receive 4 cycles of cisplatin 75mg/m2 on day 1 every 3 weeks.
Drug: placebo — Patients will receive 4 cycles of placebo IV on day 1 every 3 weeks.
  Arms: placebo group
Procedure: radical resection of esophageal carcinoma — Patients will receive radical resection of esophageal carcinoma after 4 cycles of chemotherapy.

SUMMARY:
This is a randomized, double-blind, placebo-controlled Ib/Ⅱ clinical study to evaluate the safety and effect of anti-PD-L1 antibody (ZKAB001) in neoadjuvant chemotherapy of esophageal squamous carcinoma in combination with Alb-paclitaxel and cisplatin. The immunotherapy will be given before and after the operation every three weeks.

ELIGIBILITY:
Key inclusion Criteria:

1. Aged 18 to 75 years old of either gender;
2. A histopathological diagnosis of esophageal squamous cell carcinoma with a clinical stage of T2N+M0 or T3-4aN+/-M0 according to the 8th edition of the UICC staging system;
3. ECOG score 0-1;
4. Estimated life expectancy >3 months;
5. BMI ≥18.5kg/m2 or PG-SGA score A/B;
6. The function of important organs meets the following requirements:

   1. white blood cell count (WBC) ≥ 3.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L, platelets ≥ 100×109/L, hemoglobin ≥ 90g/L;
   2. ALT, AST and AKP ≤ 2.5×ULN;
   3. serum albumin ≥ 30g/L;
   4. total bilirubin ≤ 1.5×ULN;
   5. serum creatinine ≤ 1.0×ULN, creatinine clearance rate ≥60 mL/min;
   6. INR ≤ 1.5, PT≤ 1.5×ULN;
7. Cardiac function: ≤I, pulmonary function: FEV1 >1.2L, FEV1% >40%, liver function: Child-Pugh 5-6;
8. Serum HCG negative in premenopausal women ;
9. Ability to understand the study and sign informed consent.

Key exclusion Criteria:

1. Cervical esophageal carcinoma;
2. Patients who have been treated previously with anti-tumor therapy (including chemotherapy, radiotherapy, surgery, immunotherapy, etc.);
3. Known or suspected allergy or hypersensitivity to monoclonal antibodies, any ingredients of anti-PD-L1 antibody and chemotherapeutic drugs;
4. Active autoimmune diseases;
5. A history of allogeneic stem cell transplantation and organ transplantation;
6. A history of interstitial lung disease or non-infectious pneumonia;
7. Patients who cannot tolerate chemotherapy or surgery due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia;
8. A history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases;
9. Presence of active hepatitis B (HBV DNA ≥ 200 IU/mL or 103 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay);
10. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
11. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer;
12. Lymph node metastasis in neck, supraclavicular, abdominal cavity, retroperitoneum and pelvic cavity (except paracardial and left gastric lymph nodes).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
major pathologic response rate | Two weeks after surgery.
  The rate of pathologic 1a and 1b after neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
R0 resection rate | Two weeks after surgery.
  The R0 resection rate of esophagectomy.
pathological complete response rate | Two weeks after surgery.
  The rate of pathologic 1a after neoadjuvant chemotherapy.
disease free survival | From the date of surgery until the date of death due to disease progression or the date of first documented disease progression whichever came first, assessed up to 24 months.
  The 2-year disease free survival of the whole group.
disease free survival rate | From the date of surgery until the date of death due to disease progression or the date of first documented disease progression whichever came first, assessed up to 24 months.
  The 2-year disease free survival rate of the whole group.
event free survival | From the date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
  The 2-year event free survival of the whole group.
event free survival rate | From the date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
  The 2-year event free survival rate of the whole group.
overall survival rate | From the date of randomization until the date of death from any cause or the date of last follow-up whichever came first, assessed up to 24 months.
  The 2-year overall survival rate of the whole group.
overall survival | From the date of randomization until the date of death from any cause or the date of last follow-up whichever came first, assessed up to 24 months.
  The 2-year overall survival of the whole group.
adverse events rate | From the date of randomization to 90 days after the last chemotherapy.
  The incidence rate of treatment-related adverse events of the whole group assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: SHUGENG GAO, MD, Study Director — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Kelsen DP, Ginsberg R, Pajak TF, Sheahan DG, Gunderson L, Mortimer J, Estes N, Haller DG, Ajani J, Kocha W, Minsky BD, Roth JA. Chemotherapy followed by surgery compared with surgery alone for localized esophageal cancer. N Engl J Med. 1998 Dec 31;339(27):1979-84. doi: 10.1056/NEJM199812313392704. PMID 9869669
- [Background] Lin CC, Hsu CH, Cheng JC, Wang HP, Lee JM, Yeh KH, Yang CH, Lin JT, Cheng AL, Lee YC. Concurrent chemoradiotherapy with twice weekly paclitaxel and cisplatin followed by esophagectomy for locally advanced esophageal cancer. Ann Oncol. 2007 Jan;18(1):93-98. doi: 10.1093/annonc/mdl339. Epub 2006 Oct 6. PMID 17028244
- [Background] Polee MB, Tilanus HW, Eskens FA, Hoekstra R, Van der Burg ME, Siersema PD, Stoter G, Van der Gaast A. Phase II study of neo-adjuvant chemotherapy with paclitaxel and cisplatin given every 2 weeks for patients with a resectable squamous cell carcinoma of the esophagus. Ann Oncol. 2003 Aug;14(8):1253-7. doi: 10.1093/annonc/mdg328. PMID 12881388
- [Background] Shapiro J, van Hagen P, Lingsma HF, Wijnhoven BP, Biermann K, ten Kate FJ, Steyerberg EW, van der Gaast A, van Lanschot JJ; CROSS Study Group. Prolonged time to surgery after neoadjuvant chemoradiotherapy increases histopathological response without affecting survival in patients with esophageal or junctional cancer. Ann Surg. 2014 Nov;260(5):807-13; discussion 813-4. doi: 10.1097/SLA.0000000000000966. PMID 25379852
- [Derived] Li Y, Zhou A, Liu S, He M, Chen K, Tian Z, Li Y, Qin J, Wang Z, Chen H, Tian H, Yu Y, Qu W, Xue L, He S, Wang S, Bie F, Bai G, Zhou B, Yang Z, Huang H, Fang Y, Li B, Dai X, Gao S, He J. Comparing a PD-L1 inhibitor plus chemotherapy to chemotherapy alone in neoadjuvant therapy for locally advanced ESCC: a randomized Phase II clinical trial : A randomized clinical trial of neoadjuvant therapy for ESCC. BMC Med. 2023 Mar 8;21(1):86. doi: 10.1186/s12916-023-02804-y. PMID 36882775
- See also: GLOBOCAN 2018: oesophagus cancer fact sheet — http://gco.iarc.fr/today/data/factsheets/cancers/6Oesophagus-fact-sheet.pdf.